CLINICAL TRIAL: NCT02047591
Title: Study of a Therapy Without Drugs, Supplementary to an Usual Treatment for the Pains Caused by Removing the Redon's Drain From a 7 to 17 Years Old Child in Pediatric Surgery.
Acronym: TOUTETDOU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: I11017
Record Dates: First submitted 2014-01-26; First posted 2014-01-28 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2016-02

CONDITIONS: Surgical Operation With the Settle of a Redon's Drain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Relaxing-touch method (Experimental)
  Interventions: Other: Relaxing-touch method
- Usual care (No Intervention)

INTERVENTIONS:
Other: Relaxing-touch method
  Arms: Relaxing-touch method

SUMMARY:
The 3rd governmental plan of fighting against the pain favored the development and the evaluation of the efficiency of the non pharmacological methods. Its results always showes a lack of knowledge of these methods and the utility to pursue the researches.

In the department of pediatric surgery of the university hospital of Limoges, the relaxing-touch is one of these methods which is more and more used. The healthcare staff noticed the beneficial effects of such an empirical method in terms of comfort and quality of life for the children.

In 2011, a pilot study led in this department showed that, in spite of the usual treatment, the removal of the Redon's drain remains painful for 25 % of the children (score on the pain scale > or = 4). This result convinced the medical team to write a protocol of research from the following hypothesis: the implementation of a protocol of the Redon's drain removal associated to the relaxing touch and usual treatment could lead to a decrease of the acute pain for a 7 to 17 years old child.

ELIGIBILITY:
Inclusion Criteria:

* Children > or = 7 and < 18 years old
* Hospitalization for surgery having required the settle of a Redon's drain during surgery.
* The presence of at least one of the legal representatives with the child during the care.
* The consent of at least one of the legal representatives and agreement of the child for the relaxing-touch method.
* The affiliation of one of the legal guardian to the social security.

Exclusion Criteria:

* Children with an intellectual deficiency preventing the use of the scale EVA from the pain.
* Children having already had one or several removal of the Redon's drain: the negative memory of the pain for a similar act could falsify the score of pain
* Children refusing the usual care of the pain in the department by the MEOPA.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 232 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
To compare the score of pain, just after the removal of the Redon's drain | 5 minutes
  The score of pain, just after the removal of the Redon's drain, constitutes the main end point. It will be collected by the score of the EVA (scores from 0 to 10)

SECONDARY OUTCOMES:
To compare, for 2 groups, the Score of pain: EVA scale (score 0-10). | 5 minutes
  Score of pain: EVA scale (score 0-10). The 2 groups average EVA level will be compared.
Percentage of children with a pain rating ≥ 4 | 5 minutes
  The Percentage of children with a pain rating ≥ 4 will be compared between the two groups in children aged 7 to 11 and 12 to 17 years old
To compare, for 2 groups, the average level of EVA-anxiety scores | 5 minutes
  Comparison of the average level of "EVA-anxiety" scores in the two groups of children before treatment
Proportion of children with a pain level ≥ 4 during removal of the drain | 5 minutes
  the proportion of children with a pain level ≥ 4 during removal of the drain in the group of children who underwent an orthopedic procedure; a visceral act; an act thoracic; an act for gynecomastia; an act for burn treatment by prosthesis expansion;

CONTACTS AND LOCATIONS:
Overall Officials: Laurent FOURCADE, MD, Principal Investigator — University Hospital of Limoges
Locations (1):
- Limoges Hospital, Limoges, France

REFERENCES:
- [Background] Effectiveness of pain relief by
- See also: Results of the research — https://doi.org/10.25965/reasci.152